CLINICAL TRIAL: NCT05708014
Title: Personalized Prevention for Couples
Brief Title: Personalized Prevention for Couples: A 16-month Digital RCT
Acronym: LuvHub
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R01MH126880-02 (NIH); 5R01MH126880-04 (NIH)
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hiv; HIV Infections; Sexually Transmitted Infection; Sexually Transmitted Diseases; Sexual Behavior; Risk Reduction
Keywords: Prevention; Relationship functioning; Adherence; Prevention strategies
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Sexually Transmitted Diseases; Sexual Behavior; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: 16-month randomized control trial with delayed, educational control condition of 8 months.
Who Masked: Participant
Masking Description: Participants and relationship partner will not know in advance which arm they are assigned and randomized to in the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): From baseline to 16-months, participants randomized to the intervention arm will have access to the LuvHub web app intervention and all of its contents (5 modules, resources, etc.), including post-baseline assessments that will occur every 4 months (4, 8, 12, & 16-months).
  Interventions: Behavioral: Intervention LuvHub
- Waitlist Control (Experimental): From baseline to 8-months, participants in the waitlist control condition will have access to the LuvHub web app for post-baseline assessments of 4 and 8 months, and the resources section.
  From 8-months to 16-months, participants randomized to the waitlist control arm will then have access to the LuvHub web app intervention and all of its contents (5 modules, resources, etc.), including post-baseline assessments that will occur every 4 months (12 & 16-months).
  Interventions: Behavioral: Waitlist Control LuvHub

INTERVENTIONS:
Behavioral: Intervention LuvHub — From day 1 to day 487 (i.e., entire 16-month duration, post baseline) of the trial, participants randomized to the intervention arm will have access to use the five modules as directed. The LuvHub intervention includes modules focused on topics of: HIV/STI prevention, sexual agreements, communication/decision-making skills, strengthening relationships and creating goals, and physical activity.
  Other Names: LuvHub
  Arms: Intervention
Behavioral: Waitlist Control LuvHub — From day 243 to day 487 (i.e., starting after 8-month assessment) of the trial, participants randomized to the waitlist control condition will have access to use the five modules as directed. The LuvHub intervention includes modules focused on topics of: HIV/STI prevention, sexual agreements, communication/decision-making skills, strengthening relationships and creating goals, and physical activity.
  Other Names: LuvHub
  Arms: Waitlist Control

SUMMARY:
This couples-based, digital health intervention project is serostatus neutral and seeks to determine efficacy for: a) use and adherence to evidence-based HIV/STI prevention-care strategies; b) creation and adherence to a tailored prevention-care plan; c) creation and adherence to a tailored sexual agreement; and d) improvements in other relationship dynamics among male couples who are in a relationship (defined as greater than 3 months or more).

DETAILED DESCRIPTION:
The project draws on our strong findings from the preliminary work we conducted in the US (R34 pilot randomized control trial & mixed method acceptability project). The 5-year project will revise and update an existing digital health couples-based HIV/STI prevention toolkit intervention that showed promise for reducing couples' HIV risk. The intervention is theoretically grounded in Couples Interdependence Theory for health behavior change. The project is a 16-month randomized control trial with 375 at-risk male couples using a delayed, educational control condition of 8 months. Our Specific Aims are to: 1) examine efficacy of the intervention on couples' a) formation and adherence to a risk-reduction plan and agreement, b) relationship functioning, c) self-reported and biomarker-confirmed indicators of risk (sexual behavior and STI), and engagement in HIV prevention (PrEP adherence) and care (ART adherence); 2) evaluate use of the intervention over time by using three different data sources; 3) explore moderating and mediating effects on couples' outcomes a-c. The project has high Public Health significance given the HIV disparities and the importance of attending to couples' unique relationship and prevention needs.

ELIGIBILITY:
Inclusion Criteria:

1. assigned male at birth and currently identify as male (cis-gender) or gender queer;
2. has had condomless anal sex (CAS) within the prior 3 months;
3. both partners endorse being in a relationship with one another, defined as "someone you feel emotionally or romantically committed to above all others, and may be referred to as partner, husband, boyfriend etc.";
4. be in a relationship with current partner for at least 3 months;
5. be at least 18 years of age;
6. not have any history of intimate partner violence since relationship began;
7. self-report not feeling coerced by partner to take part in the study activities,
8. has own Internet/web-connected device (e.g. smartphone, laptop, tablet, computer);
9. lives in the U.S. and plans to live in the U.S. for the next 16 months;
10. willing to complete the activities required to obtain and mail back their biomedical data (i.e., self-administer a rapid HIV test (if applicable), willing to use swabs to self-collect their own specimens for STI testing, willing to provide dried blood spot for ART adherence (if applicable), willing to provide dried blood spot for PrEP adherence (if applicable).

Exclusion Criteria:

* Does not meet one or more of the inclusion criteria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender men
Enrollment: 778 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Change in HIV incidence by comparing results from test kits received at baseline to 16-months. | Baseline to 16-months
  Participants will be asked to provide sample to test for HIV at baseline and 16-months, using at-home self-collection test kits.
  Count: New HIV and STI diagnosis via biomedical testing at follow-up occurring 16 months after baseline randomization.
Change in STI incidence by comparing results from test kits received at baseline to 16-months. | Baseline to 16-months
  Participants will be asked to provide samples to test for STIs at baseline and 16-months, using at-home self-collection test kits.
  Count: New HIV and STI diagnosis via biomedical testing at follow-up occurring 16 months after baseline randomization.
Changes in relationship communication patterns by comparing responses from baseline to 8-months, 8-months to 16-months, and baseline to 16-months. | Baseline to 8-months, 8-months to 16-months, baseline to 16-months
  Participants will be asked 11 questions with Likert-type scale responses (range 1-9) at all time points: 3 items for mutual constructive communication (MCC): higher scores represent greater MCC. 8 items for avoidance and withdrawal patterns (AW): higher scores represent greater AW.
  Changes in mean scores of MCC and AW (individual, couple), respectively, will be evaluated from baseline to 8-months, 8-months to 16-months, and baseline to 16-months.
  Heavey CL, Brandon ML, Zumtobel DC, et al. The Communication Patterns Questionnaire: The reliability and validity of a constructive communication subscale. J Marriage Fam. 1996;58(3):796-800. No PMID.
  Futris TG, Campbell K, Nielsen RB, Burwell SR. The Communication Patterns Questionnaire-Short Form: A Review and Assessment. Fam J. 2010;18(3):275-87. No PMID.
Changes in relationship commitment by comparing responses from baseline to 8-months, 8-months to 16-months, and baseline to 16-months. | Baseline to 8-months, 8-months to 16-months, baseline to 16-months
  Participants will be asked about their relationship commitment at all time points, using a validated theoretical measure containing 13 questions with Likert-type scale responses (range 1-5). Higher scores represent greater commitment to the relationship.
  Changes in mean scores (individual, couple) from baseline to 8-months, 8-months to 16-months, and baseline to 16-months.
  Rusbult CE, Martz JM, Agnew CA. The investment model scale: Measuring commitment level, satisfaction level, quality of alternatives, and investment size. Pers Relatsh. 1998;5(4):357-391. No PMID.
  Rodrigues D, Lopes D. The Investment Model Scale (IMS): further studies on construct validation and development of a shorter version (IMS-S). J Gen Psychol. 2013;140(1):16-28. PMID: 24837343.
Changes in relationship trust by comparing responses from baseline to 8-months, 8-months to 16-months, and baseline to 16-months. | Baseline to 8-months, 8-months to 16-months, baseline to 16-months
  Participants will be asked about their relationship trust at all time points, using a validated theoretical measure containing 8 questions with Likert-type scale responses (range: 0-6). Higher scores represent greater trust toward the partner in the relationship.
  Changes in mean scores (individual, couple) from baseline to 8-months, 8-months to 16-months, and baseline to 16-months.
  Larzelere RE, Huston TL. The Dyadic Trust Scale: Toward understanding interpersonal trust in close relationships. J Marriage Fam. 1980;42(3):595-604. No PMID.
Changes in relationship communal coping by comparing responses from baseline to 8-months, 8-months to 16-months, and baseline to 16-months. | Baseline to 8-months, 8-months to 16-months, baseline to 16-months
  Participants will be asked 42 items (range 1-5): outcome efficacy to reduce HIV threat subscale of joint effort (7 items), communication (7 items), and planning and decision-making (7 items); couple efficacy reduce HIV threat subscale of joint effort (7 items), communication (7 items), and planning and decision-making (7 items). Higher scores represent greater attitudes to achieve outcomes or couple's confidence that together they can engage in communal coping efforts.
  Changes in mean scores (individual, couple) from baseline to 8-months, 8-months to 16-months, and baseline to 16-months.
  Salazar LF, Stephenson RB, Sullivan PS, et al. Development and validation of HIV-related dyadic measures for men who have sex with men. J Sex Res. 2013;50(2):164-177. PMID: 22206480.
Changes in relationship transformation of motivation by comparing responses from baseline to 8-months, 8-months to 16-months, and baseline to 16-months. | Baseline to 8-months, 8-months to 16-months, baseline to 16-months
  Participants will be asked about their relationship transformation of motivation (ToM) at all time points, using 2 questions (range 1-5).
  ToM measures (1) cognitive and (2) emotional response to the health threat. Higher scores represent greater cognitive response and emotional response, respectively.
  Changes in mean scores (individual, couple) from baseline to 8-months, 8-months to 16-months, and baseline to 16-months.
  Salazar LF, Stephenson RB, Sullivan PS, et al. Development and validation of HIV-related dyadic measures for men who have sex with men. J Sex Res. 2013;50(2):164-177. PMID: 22206480.
Changes in the creation of a detailed risk reduction plan by comparing responses from baseline to 8-months, 8-months to 16-months, and baseline to 16-months. | Baseline to 8-months, 8-months to 16-months, baseline to 16-months
  Participants will be asked if they created a detailed risk-reduction plan that contains evidence-based strategies with their partner at all time points, using a dichotomous measure containing yes/no responses.
  Changes in responses (individual, couple) from baseline to 8-months, 8-months to 16-months, and baseline to 16-months.
Changes in the creation of a detailed agreement by comparing responses from baseline to 8-months, 8-months to 16-months, and baseline to 16-months. | Baseline to 8-months, 8-months to 16-months, baseline to 16-months
  Participants will be asked if they created a detailed agreement with their partner at all time points, using a dichotomous measure containing yes/no responses.
  Changes in responses (individual, couple) from baseline to 8-months, 8-months to 16-months, and baseline to 16-months.
Changes in adherence to risk-reduction plan by comparing responses from baseline to 8-months, 8-months to 16-months, and baseline to 16-months. | Baseline to 8-months, 8-months to 16-months, baseline to 16-months
  Participants will be asked whether they had adhered to their risk reduction plan at all time points.
  Changes to categorical responses (yes/no) at individual and couple levels from baseline to 8-months, 8-months to 16-months, and baseline to 16-months.
Changes in adherence to agreement by comparing responses from baseline to 8-months, 8-months to 16-months, and baseline to 16-months. | Baseline to 8-months, 8-months to 16-months, baseline to 16-months
  Participants will be asked whether they had adhered to their agreement at all time points.
  Changes to categorical responses (yes/no) at individual and couple levels from baseline to 8-months, 8-months to 16-months, and baseline to 16-months.
Changes in the number of evidence-based prevention strategies being used over time by comparing responses from baseline to 8-months, 8-months to 16-months, and baseline to 16-months. | Baseline to 8-months, 8-months to 16-months, baseline to 16-months
  Participants will be asked to select which evidence-based HIV/STI prevention strategies they are currently using at all time points.
  Changes to categorical responses (yes/no) at individual and couple levels from baseline to 8-months, 8-months to 16-months, and baseline to 16-months.

CONTACTS AND LOCATIONS:
Overall Officials: Jason W Mitchell, PhD, Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Findings from aim 1-3 will be shared via presentation(s) at peer-reviewed national and international conferences, such as the International AIDS Conference, IAS, AIDS Impact, and the International Congress of Behavioral Medicine.
  Findings resulting from the analysis of the data related to the 6-month pilot randomized control trial will be shared as Research Papers in leading, peer-reviewed journals, such as: JMIR Mhealth Uhealth, AIDS and Behavior, JAIDS, and Prevention Science.
  A de-identified version of the project's final analytic dataset and codebook will be shared and made available via a download link located at the Florida International University Digital Repository.
Time Frame: Data will become available Fall 2026.
Access Criteria: User registration will be required in order to access or download files. As part of the registration process, users must agree to the conditions of use governing access to the public release data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource.